CLINICAL TRIAL: NCT00090064
Title: Phase II Clinical Trial Testing the Safety and Efficacy of 3,4-Methylenedioxymethamphetamine (MDMA)-Assisted Psychotherapy in Subjects With Chronic Posttraumatic Stress Disorder
Brief Title: MDMA-Assisted Psychotherapy in People With Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP1
Record Dates: First submitted 2004-08-24; First posted 2004-08-25 (Estimated); Results first posted 2021-10-25 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder
Keywords: MDMA; Methylenedioxymethamphetamine; PTSD; psychotherapy; midomafetamine
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- MDMA-assisted therapy (125 mg) (Experimental): Participants will receive an initial dose of 125 mg midomafetamine HCl orally followed 2 to 2.5 hours later by a second dose of 62.5 mg midomafetamine HCl during two 8-hour long blinded therapy sessions.
  Interventions: Drug: Midomafetamine HCl; Behavioral: Therapy
- Placebo with therapy (Placebo Comparator): Participants will receive an initial dose of 125 mg placebo orally followed 2 to 2.5 hours later by a second dose of 62.5 mg placebo during two 8-hour long blinded therapy sessions.
  Interventions: Drug: Lactose placebo pill; Behavioral: Therapy

INTERVENTIONS:
Drug: Midomafetamine HCl — 125 mg of midomafetamine HCl followed by a supplemental half-dose of 62.5 mg of midomafetamine HCl
  Other Names: MDMA HCl; 3,4-methylenedioxymethamphetamine; MDMA; Midomafetamine
  Arms: MDMA-assisted therapy (125 mg)
Drug: Lactose placebo pill — 125 mg followed by a supplemental half-dose of 62.5 mg
  Other Names: Placebo
  Arms: Placebo with therapy
Behavioral: Therapy — Non-directive therapy provided by a team of two co-therapists

SUMMARY:
The goal of this clinical trial is to compare MDMA-assisted therapy to placebo with therapy in people with chronic, treatment-resistant posttraumatic stress disorder (PTSD). The main question it aims to answer is: Is there a reduction in PTSD symptoms among people given MDMA-assisted therapy compared to placebo with therapy?

Participants will receive either MDMA-assisted therapy or placebo with therapy during two blinded experimental sessions spaced three to five weeks apart. During experimental sessions, participants receive an initial dose of 125 mg of MDMA HCl, or placebo, followed by a dose of 62.5 mg of MDMA HCl, or placebo. During this treatment period, participants will also undergo non-drug preparatory psychotherapy sessions and non-drug integrative sessions.

The study will test whether MDMA-assisted therapy can be safely given to participants. Researchers will compare PTSD symptoms in the MDMA-assisted therapy group to the placebo with therapy group to see if there is a reduction in symptoms after the treatment period.

DETAILED DESCRIPTION:
This randomized, double-blind placebo-controlled pilot study assessed the safety and effectiveness of MDMA-assisted therapy among people with chronic, treatment-resistant PTSD, including veterans. Participants were assigned to receive either MDMA-assisted therapy or placebo with therapy during two blinded experimental sessions spaced three to five weeks apart during Stage 1 of the study. During these experimental sessions, participants received an initial dose of 125 mg of MDMA HCl followed by a supplemental dose of 62.5 mg of MDMA HCl, or they received initial and supplemental doses of inactive placebo. Psychotherapists and independent raters were blinded to participants' treatment conditions. This treatment period also consisted of non-drug preparatory therapy sessions and non-drug integration therapy sessions.

During Stage 2 of the study, the blind was broken and participants assigned to receive MDMA-assisted therapy in Stage 1 underwent a third open-label experimental session of MDMA-assisted therapy. Participants assigned placebo with therapy during Stage 1 who chose to enroll in Stage 2 underwent three open-label sessions of MDMA-assisted therapy. Outcome measures were administered two months after the second experimental session in Stage 1 and four to six weeks after the second MDMA-assisted therapy session in Stage 2. A final data-collection session took place at two months after the third experimental session.

The primary objective of the study was to measure change in PTSD symptoms via CAPS-IV across the study in participants receiving MDMA-assisted therapy versus placebo with therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have current PTSD (within the past 6 months) in response to crime victimization, including childhood sexual or physical abuse, or meet criteria for PTSD in response to combat;
* Have a CAPS score showing moderate to severe PTSD symptoms;
* They must either:

  1. Have had at least one unsuccessful attempt at treatment for PTSD with a SSRI and psychotherapy;
  2. Be a veteran with PTSD symptoms that have endured for no less than one year but no more than five years
* Be at least 18 years old;
* Must be generally healthy;
* Willing to remain overnight at the study site;
* Agree to have transportation home the morning after experimental sessions;
* Are willing to be contacted via telephone for all necessary telephone contacts;
* Must have a negative pregnancy test if able to bear children and agree to use an effective form of birth control;
* Are proficient in reading English;

Exclusion Criteria:

* Are pregnant or nursing, or are able to bear children and are not practicing an effective means of birth control;
* Weigh less than 50 kg or more than 105 kg;
* Are unable to give adequate informed consent;
* Prior use of "Ecstasy" (illicit drug preparations purported to contain MDMA) more than 5 times or at any time within the previous 6 months;
* Have a history of certain excluded medical disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-03-12; Primary Completion 2008-05-02 (Actual); Study Completion 2010-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mithoefer, MD, Principal Investigator — Private Practice
Locations (1):
- Offices of Michael Mithoefer MD, Mt. Pleasant, South Carolina, United States

REFERENCES:
- [Result] Mithoefer MC, Wagner MT, Mithoefer AT, Jerome L, Doblin R. The safety and efficacy of +/-3,4-methylenedioxymethamphetamine-assisted psychotherapy in subjects with chronic, treatment-resistant posttraumatic stress disorder: the first randomized controlled pilot study. J Psychopharmacol. 2011 Apr;25(4):439-52. doi: 10.1177/0269881110378371. Epub 2010 Jul 19. PMID 20643699
- [Result] Mithoefer MC, Wagner MT, Mithoefer AT, Jerome L, Martin SF, Yazar-Klosinski B, Michel Y, Brewerton TD, Doblin R. Durability of improvement in post-traumatic stress disorder symptoms and absence of harmful effects or drug dependency after 3,4-methylenedioxymethamphetamine-assisted psychotherapy: a prospective long-term follow-up study. J Psychopharmacol. 2013 Jan;27(1):28-39. doi: 10.1177/0269881112456611. Epub 2012 Nov 20. PMID 23172889
- [Derived] Zeifman RJ, Kettner H, Ross S, Weiss B, Mithoefer MC, Mithoefer AT, Wagner AC. Preliminary evidence for the importance of therapeutic alliance in MDMA-assisted psychotherapy for posttraumatic stress disorder. Eur J Psychotraumatol. 2024;15(1):2297536. doi: 10.1080/20008066.2023.2297536. Epub 2024 Jan 4. PMID 38174611
- [Derived] Jerome L, Feduccia AA, Wang JB, Hamilton S, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. Long-term follow-up outcomes of MDMA-assisted psychotherapy for treatment of PTSD: a longitudinal pooled analysis of six phase 2 trials. Psychopharmacology (Berl). 2020 Aug;237(8):2485-2497. doi: 10.1007/s00213-020-05548-2. Epub 2020 Jun 4. PMID 32500209
- [Derived] Feduccia AA, Jerome L, Yazar-Klosinski B, Emerson A, Mithoefer MC, Doblin R. Breakthrough for Trauma Treatment: Safety and Efficacy of MDMA-Assisted Psychotherapy Compared to Paroxetine and Sertraline. Front Psychiatry. 2019 Sep 12;10:650. doi: 10.3389/fpsyt.2019.00650. eCollection 2019. PMID 31572236
- [Derived] Mithoefer MC, Feduccia AA, Jerome L, Mithoefer A, Wagner M, Walsh Z, Hamilton S, Yazar-Klosinski B, Emerson A, Doblin R. MDMA-assisted psychotherapy for treatment of PTSD: study design and rationale for phase 3 trials based on pooled analysis of six phase 2 randomized controlled trials. Psychopharmacology (Berl). 2019 Sep;236(9):2735-2745. doi: 10.1007/s00213-019-05249-5. Epub 2019 May 7. PMID 31065731

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via letters to psychotherapists and internet advertisements.
Groups:
- MDMA-assisted Therapy: Participants will receive 125 mg MDMA followed 2 to 2.5 hours later by 62.5 mg MDMA during two 8-hour long blinded therapy sessions.
Period: Overall Study
Arm/Group | MDMA-assisted Therapy | Placebo With Therapy
Started | 15 | 8
Completed | 13 | 8
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MDMA-assisted Therapy | Placebo With Therapy | Total
Number analyzed (Participants) | 15 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (7.4) | 40.8 (7.0) | 40.6 (70.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 14 | 8 | 22
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician-Administered PTSD Scale (CAPS-IV) From Baseline to 2-month Follow-up
Description: The Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-IV. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Baseline to 2 months post second experimental session
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- MDMA-assisted Therapy: Participants will receive an initial dose of 125 mg MDMA orally followed 2 to 2.5 hours later by a second dose of 62.5 mg MDMA during two 8-hour long blinded therapy sessions.
  3,4-methylenedioxymethamphetamine: 125 mg MDMA followed by a supplemental half-dose of 62.5 mg MDMA
  Therapy: Non-directive therapy provided by a team of two co-therapists
- Placebo With Therapy: Participants will receive an initial dose of 125 mg placebo orally followed 2 to 2.5 hours later by a second dose of 62.5 mg placebo during two 8-hour long blinded therapy sessions.
  Lactose placebo pill: 125 mg placebo followed by a supplemental half-dose of 62.5 mg placebo
  Therapy: Non-directive therapy provided by a team of two co-therapists
Arm/Group | MDMA-assisted Therapy | Placebo With Therapy
Number analyzed (Participants) | 12 | 8
score on a scale | -55.2 (33.54) | -20.5 (20.47)

2. Secondary Outcome: Change in Impact of Events Scale Revised (IES-R) From Baseline to 2-month Follow-up
Description: The Impact of Events Scale Revised (IES-R) is a 22-item self-report measure (for DSM-IV) designed to measure the extent to which a given stressful life event produces subjective distress. Each item corresponds directly to 14 of the 17 DSM-IV symptoms of PTSD and is rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely") for the extent to which the item was true for the participant during the past seven days. The IES-R yields a total score ranging from 0 to 88 with higher scores indicated greater distress.
Time Frame: Baseline to 2 months post second experimental session
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MDMA-assisted Therapy | Placebo With Therapy
Number analyzed (Participants) | 13 | 7
score on a scale | -29.7 (21.3) | -12.9 (15.00)

ADVERSE EVENTS:
Time Frame: On or after first day of study intervention through to follow-up visit (approximately 7 months)
Groups:
- SRRs: MDMA-assisted Therapy; SRRs: Placebo With Therapy: Spontaneously reported reactions (SRRs) collected on the day of experimental sessions and 7 days after.
Arm/Group | MDMA-assisted Therapy | Placebo With Therapy | SRRs: MDMA-assisted Therapy | SRRs: Placebo With Therapy
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/8 | 0/15 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/15 | 0/8 | 0/15 | 0/8
Other Adverse Events (participants affected / at risk) | 13/15 | 8/8 | 15/15 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MDMA-assisted Therapy (N=15) | Placebo With Therapy (N=8) | SRRs: MDMA-assisted Therapy (N=15) | SRRs: Placebo With Therapy (N=8)
Clavicle fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Syncope (Nervous system disorders) | 1 | 0 | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | MDMA-assisted Therapy (N=15) | Placebo With Therapy (N=8) | SRRs: MDMA-assisted Therapy (N=15) | SRRs: Placebo With Therapy (N=8)
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 4 | 14/14 | 8
Asthenia (General disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Bruxism (Psychiatric disorders) | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 1 | 0 | 0
Derealisation (Psychiatric disorders) | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Dissociation (Psychiatric disorders) | 1 | 0 | 0 | 0
Disturbance in attention (Psychiatric disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 8/14 | 6
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 2 | 14 | 8
Feeling hot (General disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 13/14 | 8
Hypoaesthesia facial (Nervous system disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Irritability (General disorders) | 2 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Muscle strain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 11 | 6/7
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Oropharyngeal blistering (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 3 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Sinus headache (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 2 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 12/13 | 8
Memory impairment (Psychiatric disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Flashback (Psychiatric disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Clavicle fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Difficulty Concentrating (General disorders) | 0 | 0 | 7/11 | 4/7
Drowsiness (General disorders) | 0 | 0 | 2/12 | 3/6
Dry mouth (General disorders) | 0 | 0 | 4/14 | 5
Fatigue (General disorders) | 0 | 0 | 14 | 8
Heavy legs (General disorders) | 0 | 0 | 2/11 | 0/5
Impaired gate/balance (General disorders) | 0 | 0 | 6/14 | 4/7
Increased irritability (General disorders) | 0 | 0 | 8/12 | 7
Increased private worries (General disorders) | 0 | 0 | 5/11 | 3/7
Jaw clenching, tight jaw (General disorders) | 0 | 0 | 12/14 | 6
Lack of appetite (General disorders) | 0 | 0 | 10/14 | 6
Low mood (General disorders) | 0 | 0 | 8/13 | 6
Nausea (General disorders) | 0 | 0 | 11 | 6/7
Need more sleep (General disorders) | 0 | 0 | 4/12 | 5/7
Nystagmus (General disorders) | 0 | 0 | 3/13 | 2/7
Parasthesias (General disorders) | 0 | 0 | 3/12 | 1/6
Perspiration (General disorders) | 0 | 0 | 3/13 | 6
Restlessness (General disorders) | 0 | 0 | 5/11 | 4
Sensitivity to cold (General disorders) | 0 | 0 | 10/14 | 6
Thirst (General disorders) | 0 | 0 | 2/11 | 4
Weakness (General disorders) | 0 | 0 | 5/12 | 4/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2009-01-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT00090064/Prot_005.pdf
  • Statistical Analysis Plan (2011-11-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT00090064/SAP_004.pdf